CLINICAL TRIAL: NCT02410746
Title: A Prospective, Randomised Double Blinded Study Comparing a Pectoral Nerve Block With Non-targeted Local Anaesthetic in Bilateral Breast Surgery
Brief Title: Nerve Block Versus Non-targeted Local Anaesthesia in Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BMI Healthcare (Other)
Responsible Party: Principal Investigator, Anne Dancey, Consultant Plastic Surgeon, BMI Healthcare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PECBLOCKV1
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Pain, Post Operative
Keywords: pain; surgery
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Morphine; Acetaminophen; Ibuprofen; Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard chirocaine infiltration (Active Comparator): non-targeted infiltration of 10ml 0.25% Chirocaine into breast pocket
  Interventions: Other: standard chirocaine infiltration; Other: standard post-operative analgesia
- targeted chirocaine pec block (Experimental): pectoral muscle block with 10ml 0.25% chirocaine
  Interventions: Other: targeted chirocaine pec block; Other: standard post-operative analgesia

INTERVENTIONS:
Other: targeted chirocaine pec block — 10ml 0.25% chirocaine in a specifically targeted in a nerve block
  Other Names: Pectoral nerve block
  Arms: targeted chirocaine pec block
Other: standard chirocaine infiltration — 10ml 0.25% chirocaine is infiltrated into breast pocket in a non targeted fashion
  Other Names: intra-operative analgesia
  Arms: standard chirocaine infiltration
Other: standard post-operative analgesia — A dose of morphine 0.1mg/kg will be given intra-operatively. Thereafter morphine 0.1mg/kg will be given for breakthrough pain. Patients will be prescribed regular paracetamol and ibuprofen.
  Other Names: Morphine, Paracetamol, ibuprofen, analgesia

SUMMARY:
Effective postoperative pain control is an essential component of surgery. Adequate analgesia improves patient comfort and satisfaction, thereby permitting earlier mobilisation, faster recovery and less likelihood of complications.The majority of surgeons will place 10ml of local anaesthetic into the breast pocket or inject it into the breast skin following breast surgery. A more specific technique is to identify the nerves supplying the breast and put the local anaesthetic directly around them (Pec block). This nerve block has recently been described and is increasingly being used by anaesthetists for surgery under local anaesthetic or for post-operative analgesia. It has been shown to provide better and more specific pain relief in several studies.

Anaesthetists use an ultrasound machine to identify the anatomical landmarks for the nerves and they inject into the vicinity. They do not have direct vision and there is a risk of causing morbidity or the block not being effective. It is much easier for a surgeon to apply the block, as they can see the anatomical landmarks. Despite this, very few surgeons are aware of the technique.

The study group consists of patients undergoing bilateral cosmetic breast surgery at BMI Edgbaston and Priory hospitals and Spire Parkway and Southbank hospitals in Birmingham and Worcester. If a patient consents to being involved in the research, they will have one breast randomised to receiving a pec block and the contralateral (opposite) breast will receive the same amount of local anaesthetic placed in the breast pocket in a non-targeted fashion. The patients and researcher will be blinded as to the allocation. Patients will complete a verbal numeric pain score for each breast at set intervals until they are discharged.In addition, the investigators will specifically ask which breast is the most painful at each time point.

The results of the study may improve patient care.

DETAILED DESCRIPTION:
The investigators' intention is to randomise all patients undergoing bilateral breast surgery into receiving a specific pec block in one breast and a standard infiltration of non targeted anaesthesia into the other breast. 10ml 0.25% Chirocaine will be used for each breast.

All patients attending the plastic surgery clinic at BMI Edgbaston, BMI Priory, Spire Parkway and Spire Southbank and requesting bilateral breast surgery will be approached to take part in the study. They will be given information to take home and an opportunity to ask any questions about the study.

All consenting patients who meet the inclusion criteria will have one breast randomised into a study group (pec block) and the other into a control group (standard local anaesthetic infiltration). Patients will be randomised by a computer generated code. The patient and researcher will be blinded. By necessity, the surgeon will be aware of the randomisation but will have no involvement in data collection or analysis of results.

Both groups will receive standard post-operative care and follow up. A dose of morphine 0.1mg/kg will be given intra-operatively. Thereafter morphine 0.1mg/kg will be given for breakthrough pain. Patients will be prescribed regular paracetamol and ibuprofen. The investigators will prospectively record post operative pain as rated by a verbal numerical rating scale at 0, 3, 6, 9 and 12 hours post-operatively and at 24 hours. In addition the investigators will record which breast the patient indicates is the most painful and any post-operative complications throughout the study period . The expected recruitment period is six months.

If patients consent to inclusion in the study they will sign a consent form at a second appointment or on the day of surgery. The ward and recovery nurses already have experience in administering a VNRS for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patient requesting a bilateral breast procedure (reduction, mastopexy or augmentation).
* Patient willing to sign the informed consent form agreeing to its items after explanation of the study by the operating surgeon.

Exclusion Criteria:

* Declining to give written consent.
* History of allergy to chirocaine local anaesthetic.
* Prior breast surgery.
* Chronic pain disorder.
* Significant medical co-morbidities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
targeted question as to which breast is more painful | 3 hours post-operatively
  patient is asked which breast is more painful

SECONDARY OUTCOMES:
verbal numeric rating scale(VNRS) | 3 hours post-operatively
  standard validated pain score

CONTACTS AND LOCATIONS:
Overall Officials: anne dancey, MBChB(hons), Principal Investigator — AAS
Locations (1):
- Edgbaston BMI Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
yes on individual request of the patient when study is completed